CLINICAL TRIAL: NCT03773484
Title: Application of Economics & Social Psychology to Improve Opioid Prescribing Safety (AESOPS): R21 Pilot Phase
Acronym: AESOPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Northwestern University (Other); AltaMed Health Services Corporation (Other); The Children's Clinic (Other)
Responsible Party: Principal Investigator, Jason Doctor, Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HS-CG-17-00019; R21AG057395-01 (NIH)
Record Dates: First submitted 2018-12-10; First posted 2018-12-12 (Actual); Results first posted 2022-08-16 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Opioid Use, Unspecified
Keywords: Opioids; Behavioral Research

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical Decision Support (Experimental): Clinical decision support nudges within the electronic health record to discourage unnecessary opioid prescribing through the application of "behavioral insights"-empirically-tested social and psychological interventions that affect choice. Participating clinicians will receive any of three nudges when eligibility criteria are met within a patient's chart.
  Interventions: Behavioral: Opioid naive; Behavioral: At-risk for long term use; Behavioral: Long-term opioid recipient

INTERVENTIONS:
Behavioral: Opioid naive — Visit where the order is for an included opioid and there is no prior opioid prescription with a start date of greater than 1 day and less than 91 days
Behavioral: At-risk for long term use — Visit where the order is for an included opioid, there is a prior opioid prescription with a start date greater than 1 day and less than 91 days, and there is no prior opioid prescription with a start date greater than 90 days
Behavioral: Long-term opioid recipient — Total opioid doses are at least 50 MME per day, there are two or more prior opioid prescriptions with two different start dates both greater than 1 day and less than 91 days, and there is a prior opioid prescription with a start date greater than 90 days and less than 181 days

SUMMARY:
There is a lack of evidence that long-term opioid use offers benefit for noncancer pain and an abundance of evidence of harm. The objective of the R21 pilot phase of the Application of Economics & Social psychology to improve Opioid Prescribing Safety (AESOPS) is to develop and test novel behavioral nudges to encourage adherence to pain and CDC guidelines for opioid prescribing for persons with noncancer pain. Interventions will leverage the electronic health record (EHR) to discourage unnecessary opioid prescribing through the application of "behavioral insights"-empirically-tested social and psychological interventions that affect choice.

DETAILED DESCRIPTION:
There is a lack of evidence that long-term opioid use offers benefit for noncancer pain and an abundance of evidence of harm. In 2017, the Centers for Disease Control and Prevention (CDC) issued the "CDC Guideline for Prescribing Opioids for Chronic Pain" to encourage safe and effective alternatives to opioids, discontinuation of opioids when patients do not resume normal activities and prudent dosing strategies. However, poor guideline adherence is a general concern and may impede uptake. Our prior studies have used insights from behavioral economics and social psychology to increase guideline adherence. The objective of the R21 pilot phase of the Application of Economics & Social psychology to improve Opioid Prescribing Safety (AESOPS) is to develop and test novel behavioral nudges to encourage adherence to pain and CDC guidelines for opioid prescribing for persons with noncancer pain. At the time of opioid prescribing, clinicians will be prompted with an EHR nudge when the prescribing history for the patient falls into one of the following three mutually exclusive categories: Opioid naïve, At-risk for long term use, or Long-term opioid recipient. The primary outcome is average weekly morphine milligram equivalents (MME) prescribed per-clinician.

ELIGIBILITY:
Inclusion Criteria:

* NM clinic that sees patients ≥ 18 years old whose leadership agrees to participate

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason N Doctor, PhD, Principal Investigator — University of Southern California
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Background] Kelley MA, Persell SD, Linder JA, Friedberg MW, Meeker D, Fox CR, Goldstein NJ, Knight TK, Zein D, Rowe TA, Sullivan MD, Doctor JN. The protocol of the Application of Economics & Social psychology to improve Opioid Prescribing Safety Trial 1 (AESOPS-1): Electronic health record nudges. Contemp Clin Trials. 2021 Apr;103:106329. doi: 10.1016/j.cct.2021.106329. Epub 2021 Feb 24. PMID 33636344

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 41 primary care clinicians from 3 clinics at Northwestern Medicine in Chicago, Illinois were enrolled.
Pre-assignment Details: Only clinicians listed as a treating member of the clinic receive the intervention.
Groups:
- Clinical Decision Support Nudges: 1. Opioid naïve: Visit where the order is for an included opioid and there is no prior opioid prescription with a start date of greater than 1 day and less than 91 days
  2. At-risk for long term use: Visit where the order is for an included opioid, there is a prior opioid prescription with a start date greater than 1 day and less than 91 days, and there is no prior opioid prescription with a start date greater than 90 days
  3. Long-term opioid recipient: Total opioid doses are at least 50 MME per day, there are two or more prior opioid prescriptions with two different start dates both greater than 1 day and less than 91 days, and there is a prior opioid prescription with a start date greater than 90 days and less than 181 days
Period: Pre-intervention
Arm/Group | Clinical Decision Support Nudges
Started | 41
Completed | 41
Not Completed | 0
Period: Post-intervention
Arm/Group | Clinical Decision Support Nudges
Started | 41
Completed | 36
Not Completed | 5
Not completed — 5 clinicians were excluded from analysis due to lack of prescribing data | 5

BASELINE CHARACTERISTICS:
Population: 41 clinicians from 3 Northwestern Medicine clinics were enrolled
Groups:
- Clinical Decision Support: Participating clinicians will receive any of three clinical decision support nudges within the electronic health record when eligibility criteria are met within a patient's chart:
  Opioid naïve: Visit where the order is for an included opioid and there is no prior opioid prescription with a start date of greater than 1 day and less than 91 days
  At risk for long term use: Visit where the order is for an included opioid, there is a prior opioid prescription with a start date greater than 1 day and less than 91 days, and there is no prior opioid prescription with a start date greater than 90 days
  Long term opioid recipient: Total opioid doses are at least 50 MME per day, there are two or more prior opioid prescriptions with two different start dates both greater than 1 day and less than 91 days, and there is a prior opioid prescription with a start date greater than 90 days and less than 181 days
Arm/Group | Clinical Decision Support
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 41
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 41
Average weekly milligram morphine equivalent (MME) [Mean (Standard Deviation); unit: Weekly MME]
  Opioid naive | 34.88 (86.07)
  At risk for long term use | 34.44 (168.03)

OUTCOME MEASURES:

1. Primary Outcome: Average Weekly Milligram Morphine Equivalent (MME)
Description: Average per-clinician weekly milligram morphine equivalent (MME) in the 34-week period post-intervention
Time Frame: 34 weeks
Population: Of the 41 clinicians enrolled in the study, 5 were excluded due to lack of prescribing information.
Measure: Mean (Standard Deviation); unit: Weekly MME per clinician
Groups:
- Clinical Decision Support Nudges: 1. Opioid naïve
  2. At-risk for long term use
  3. Long-term opioid recipient
  Details can be found in the Arms and Interventions section.
Arm/Group | Clinical Decision Support Nudges
Number analyzed (Participants) | 36
Weekly MME per clinician
  Opioid naïve | 34.62 (97.13)
  At-risk for long term use | 22.37 (102.67)
  Long-term opioid recipient | NA (NA) — MME cannot be calculated because the algorithm for long term opioids was not fully built at the conclusion of the study pilot. It was built and deployed for our full RCT (NCT04477304)
Statistical Analysis 1: Comparison: Clinical Decision Support Nudges; Pre post comparison for Opioid Naïve patients; Test type: Other; p = 0.43, Mixed Models Analysis; Slope = -0.008, 95% CI 2-sided [-0.03 to 0.01], Standard Error of Mean 0.011
Statistical Analysis 2: Comparison: Clinical Decision Support Nudges; Pre-post comparison for at-risk for long term use patients; Test type: Other; p = 0.24, Mixed Models Analysis; Slope = -0.019, 95% CI 2-sided [-0.051 to 0.013], Standard Error of Mean 0.016

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Clinical Decision Support Nudges
All-Cause Mortality (participants affected / at risk) | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41
Other Adverse Events (participants affected / at risk) | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/84/NCT03773484/Prot_SAP_000.pdf